CLINICAL TRIAL: NCT06145191
Title: Prophylactic Tranexamic Acid Versus Adrenaline for Bleeding Prevention During Flexible Bronchoscopy: a Double Blind, Randomized Controlled Trial
Brief Title: Prophylactic Tranexamic Acid Versus Adrenaline During Flexible Bronchoscopy
Acronym: TAVA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Goran Glodić, MD, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8.1-23/278-2; 02/013AG
Record Dates: First submitted 2023-11-13; First posted 2023-11-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Bleeding; Hemoptysis
Keywords: Bronchoscopy; Tranexamic acid; Adrenaline; Prophylaxis
MeSH Terms: conditions — Hemorrhage; Hemoptysis | interventions — Tranexamic Acid; Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multiple arm randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic acid
- Adrenaline (Experimental)
  Interventions: Drug: Adrenaline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Prophylactic topical application (1x) of tranexamic acid (100mg, 2ml, room temperature) before sampling
  Arms: Tranexamic acid
Drug: Adrenaline — Prophylactic topical application (1x) of adrenaline (1:10.000, 2ml, room temperature) before sampling
  Arms: Adrenaline
Drug: Placebo — Prophylactic topical application (1x) of placebo (0.9% NaCl, 2ml, room temperature) applied before sampling
  Other Names: 0.9% NaCl
  Arms: Placebo

SUMMARY:
Endobronchial bleeding is a common complication of bronchoscopy. Major bleeding, although rare, can be life threatening and often requires advanced therapeutic interventional pulmonary procedures which are not widely available. Minor bleeding can negatively impact outcomes such as diagnostic yield, sample size and bronchoscopy duration. Both adrenaline and tranexamic acid are successfully used topically for hemostasis during diagnostic bronchoscopy. The aim of this study is to evaluate the efficacy of prophylactically applied adrenaline and tranexamic acid in bleeding prevention during diagnostic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing diagnostic bronchoscopy with sampling (including transbronchial biopsy, endobronchial forceps biopsy, brushing, transbronchial needle aspiration)
* Signed informed consent

Exclusion Criteria:

* Any existing contraindication for diagnostic bronchoscopy
* Coagulopathy (PV INR > 1.3)
* Thrombocytopenia (<50x10*9 or anemia (Hgb <80 g/L)
* DOAC, LMWH or antiplatelet drug therapy
* Thrombophilia, history of pulmonary embolism or deep vein thrombosis
* Contraindication for endobronchial application of adrenaline
* Uncontrolled coronary artery disease, cerebrovascular disease or arrhythmia
* Uncontrolled pulmonary hypertension
* Cardiovascular decompensation
* Severe hypoxia (PaO2 <60mmHg, SaO2 <90% with an FiO2 >=60%)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Number (N) of bleeding episodes / bleeding rate (%) in each group | through study completion, an average of 1.5 years
  Number of clinically relevant bleeding episodes after prophylactic application of tranexamic acid, adrenaline and placebo (0.9% NaCl)

SECONDARY OUTCOMES:
Severity of bleeding after prophylaxis | through study completion, an average of 1.5 years
  Mean severity of bleeding assessed by a visual analogue scale (VAS; 1 minor bleeding - 10 major life threatening bleeding) by the operating bronchoscopist in each group
Number (N) of drug applications needed for bleeding control | through study completion, an average of 1.5 years
  Number (N) of drug applications needed for bleeding control in each group if bleeding occured despite prophylaxis
Number (N) of bleeding episodes / bleeding rate (%) in each group stratified according to sampling type and indication | through study completion, an average of 1.5 years
  Bleeding rate in different subgroups of patients (i.e. TBNA, forceps biopsy, brush)
Number (N) of samples taken in each group | through study completion, an average of 1.5 years
  Mean total number (N) of samples taken in each group
Adverse events | through study completion, an average of 1.5 years
  Number (N) of adverse events in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No